CLINICAL TRIAL: NCT05459792
Title: Comparative Study Between the Effect of Ultrasound Guided Median Nerve Block , Radial Nerve Block and Local Infiltration on Feasibility of Radial Artery Cannulation in Patients Undergoing Major Surgeries. A Randomized Control Study
Brief Title: Comparative Study Between the Effect of Ultrasound Guided Median Nerve Block , Radial Nerve Block and Local Infiltration on Feasibility of Radial Artery Cannulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed nabih youssef, Lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-52-2022
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Radial Artery Cannulation
MeSH Terms: interventions — Anesthesia, Local; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done by computer generated numbers and concealed by serially numbered, opague and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside. This study will be performed by 2 anaesthetists; one anaesthetist who is experienced in performing the blocks will be allocated to perform either the median or radial or local infiltration according to a computer-generated sequence of random numbers and sealed envelope, and the other anesthetist who is experienced in performing ultrasound examinations and radial cannulation, will be blinded to the technique performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ultrasound guided median nerve block (Experimental): A linear transducer will be placed on the ventral aspect of the mid-forearm, where the median nerve is visible in the fascial plane between the flexor digitorum superficialis and flexor digitorum profundus after raising a skin wheal using local anesthetic, the needle will be introduced in-plane view from lateral to medial and aimed at the fascial plane adjacent to the median nerve.
  Interventions: Procedure: median nerve block
- ultrasound guided radial nerve block (Experimental): A linear transducer will be placed on the forearm: at the elbow (the radial nerve between the brachioradialis and the biceps muscle). the preferred approach is to start proximally above the elbow and identify the radial nerve as a triangular hyperechoic structure coming off the distal humerus. then following this distally to the antecubital fossa, where the nerve will branch into its superficial and deep branches. the needle will be introduced in-plane view from lateral to medial aimed at the fascial plane adjacent to the radial nerve.
  Interventions: Procedure: radial nerve block
- local infiltration (Placebo Comparator): Intradermal infiltration followed by a subcutaneous injection with a total of 3 mL of 0.25% bupivacaine with1% lidocaine with a27- G needle.
  Interventions: Procedure: local infiltration

INTERVENTIONS:
Procedure: median nerve block — It will be given by one researcher using 5 ml 0.25% bupivacaine with 1% lidocaine for each nerve block after negative aspiration for blood so as to cover the nerve circumferentially
  Other Names: peripheral nerve block
  Arms: ultrasound guided median nerve block
Procedure: radial nerve block — It will be given by one researcher using 5 ml 0.25% bupivacaine with 1% lidocaine for each nerve block after negative aspiration for blood so as to cover the nerve circumferentially
  Other Names: peripheral nerve block
  Arms: ultrasound guided radial nerve block
Procedure: local infiltration — intradermal infiltration followed by a subcutaneous injection with a total of 3 mL of 0.25% bupivacaine with1% lidocaine with a27- G needle
  Other Names: bupivacaine and lidocaine infiltration
  Arms: local infiltration

SUMMARY:
Arterial line placement is often needed in various critical care settings. It is a basic procedure performed for continuous blood pressure (BP) monitoring and rapid access for repeated arterial blood gas samples, as it is considered to be more precise than measurement of BP by other noninvasive devices, especially in the critically ill patients or those on continuous infusions of vasoactive drugs.Arterial line placement is presumed to be a relatively safe procedure, with a rate of major complications that is below 1%. The most common site of cannulation is the radial artery, primarily due to the ease of access owing to the superficial nature of the vessel and the ease with which the site can be maintained. Additional advantages of radial artery cannulation include anatomical reliability and the less complications. However placement of a radial artery catheter can, at times, be difficult because many patients who emergently need a catheter may have a weak arterial pulse due to dehydration or blood loss or may have some form of peripheral vascular disease. Although it is usually a well-tolerated procedure, it is considered more painful than intravenous (i.v.) cannula placement, particularly in case of multiple attempts of cannulation

In this study the investigators will assess the effect of ultrasound guided median nerve block, radial nerve block and local infiltration with lidocaine on feasibility of radial artery cannulation in patients undergoing major surgeries

Objectives

1. To evaluate the effect of ultrasound guided median nerve block, radial nerve block and local infiltration on feasibility of radial artery cannulation
2. To determine the effect of ultrasound guided median nerve block, radial nerve block and local infiltration in reducing discomfort and complicationassociated with radial arterial cannulation .

3. To evaluate the effect of ultrasound guided median nerve block, radial nerve block and local infiltration in radial artery diameter and blood flow for radial arterial cannulation

DETAILED DESCRIPTION:
This a randomized control trial is designed to include (126) patients ASA physical status II patients ranging from(18) to(70)years old scheduled for elective surgery who required arterial cannulation prior to the induction of general anesthesia.

Patients meeting the inclusion criteria will be randomly assigned to receive either :

Group I :median nerve block technique (n=42) GroupII: radial nerve block technique:(n=42) Group III:local infiltrationtechnique(n=42)

Anesthesia management After arrival to the anaesthetic room, An 18-gauge intravenous cannula will be placed at the forearm on the opposite arm, standard monitoring will be used (non-invasive arterial blood pressure, ECG, pulse oximetry) Parameters like heart rate and mean blood pressure will be recorded at baseline and after 15 min of the block. Premedication will be given intravenously in the form of 0.03 mg/kg midazolam The patient will be in a supine position with the operative arm abducted to 90 and supported on an arm board .

An ultrasound device with a high-frequency linear array probe( siemens acuson x 300 ultrasound with 8-14 MHz) will be used for the measurement of the transverse diameter and peak velocity of the radial artery. The high frequency probe will be kept transeversaly on the radial artery, 1 cm proximal to the radial styloid process.The diameter of the radial artery will be measured as the horizontal distance between the 2 inner walls of the artery using the electronic calliper in the US machine,Transverse diameters will be measured by M-mode ultrasound, and the M mode sample line will always be adjusted to pass through the center of vessels to measure the diameters more precisely. All peak velocities will be measured using the pulsed-wave Doppler ultrasound mode. The Doppler sampling volume will be placed in the center of the blood vessel, and the width of the sampling range gate is 2 mm. Doppler angle correction will be performed when measuring velocity, with the calibration main line parallel to the direction of blood flow and at an angle of 50-60°.this measurment will be noted at baseline and 5 min after successful block or local infilitration, every 30 minutes intraoperative, and every 4 hours for the first 24 hours or till radial cannula is removed which ever is sooner.

Nerve blocks:

the various nerves will be visualised and blocked using 22 G 50 mm insulated nerve Sonoplex needle. All blocks will be given by one researcher using 5 ml 0.25% bupivacaine with 1% lidocaine for each nerve block after negative aspiration for blood so as to cover the nerve circumferentially The various locations of the nerve blocks will be:

1. Radial nerve: in the forearm: at the elbow (the radial nerve between the brachioradialis and the biceps muscle). the preferred approach is to start proximally above the elbow and identify the radial nerve as a triangular hyperechoic structure coming off the distal humerus. then following this distally to the antecubital fossa, where the nerve will branch into its superficial and deep branches . the needle will be introduced in-plane view from lateral to medial aimed at the fascial plane adjacent to the radial nerve.
2. Median nerve: Mid forearm (between the superficial and deep compartment) A linear transducer will be placed on the ventral aspect of the mid-forearm, where the median nerve is visible in the fascial plane between the flexor digitorum superficialis and flexor digitorum profundus after raising a skin wheal using local anesthetic, the needle will be introduced in-plane view from lateral to medial and aimed at the fascial plane adjacent to the median nerve.

local infiltration: Patients in this group received an intradermal infiltration followed by a subcutaneous injection with a total of 3 mL of 0.25% bupivacaine with1% lidocaine with a27- G needle.

Sensory blockade of the median, radial nerves will be graded according to the previously validated 3point scale using a cold test: respectively: 0 = no perception, 1 = decreased sensation, or 2 = normal sensation. it will be measured every 5 min . Blocks will be assumed to be successful if there is absence of sensation to ice (sensory block score = 0) If complete sensory blockade will not be achieved within 30 minutes, the affected subject will be excluded from the study and categorized as a block failure.

The operator will reassess the radial pulse and will grade the change in palpability of radial pulse from 0 to 4 as follows:

Grade 0 : radial pulse not palpable after the injection. Grade 1 : radial pulse become feeble after the injection Grade 2: palpability of radial pulse remains the same after the injection Grade 3: radial pulse become better palpable after the injection Grade 4 : radial pulse become bounding after the injection

Arterial cannulation will be intended to be performed after varification of successful blocks or local infiltiration, the arm will be abducted at an angle of 70 to 90 and the wrist will be hyper extended to facilitate palpation and cannulation of the radial artery. After identification of the optimal site for cannulation of the radial artery, the overlying skin will be disinfected with a swab impregnated with an alcohol- based skin disinfectant solution.

An arterial line will be then placed in the usual fashion using a standard Arrow kit, which will conclude the subject's participation in this study. The start time will be defined as the initial needle penetration through the skin. The time to successful arterial cannulation will be measured as removal of the metal needle and continuation of a flash of arterial blood. Failure to cannulate will be quantified as numbers of needle tips completely withdrawn from the skin . The success rate will be defined as successful cannulation of the radial artery in 3 attempts or fewer.

Patients will be asked to rate their discomfort using a number from 0 meaning no discomfort to 10 meaning strongest imaginable discomfort." In case of an unsuccessful cannulation or a failure cannulation will be started at an alternative site. Further cannulation attempts at an alternative site will not be assessed.

Post cannulation complication will be recorded such as arterial spasm, ischemia, thrombosis and hematoma formation.

Measurement tools

1. Patients demographic data will be collected; age, gender, weight, type of surgery and duration of surgery.
2. The ultrasound measurements (The peak velocity (mm/s)and transverse diameter(mm) values of radial artery at base line , 5 min after successful blocks or local infilitration, every 30 minutes intra operative, and every 4 hours for the first 24 hours or till radial cannula is removed which ever is sooner.

3 -Parameters like heart rate and mean blood pressure will be recorded at baseline and 5 min after successful blocks or local infilitration, every 30 minutes intraoperative.

4- feasability of cannulation: defined as number of attempts of cannulation, and time taken in seconds till successful cannulation.

5- Incidence of post cannulation complication such as arterial spasm , ischemia ,thrombosis and hematoma formation in the first 24 hours postoperative.

6- The degree of palpability of radial pulse

ELIGIBILITY:
Inclusion Criteria:

1. Gender both males and females
2. ASA Class II
3. Age 18-70 years
4. Patients undergoing surgeries requiring radial arterial cannulation expected to be needed , and in place for the first 24 hours postoperatively as thoracic surgeries(e,g lobectomy, pneumonectomy),major vascular surgeries (carotid end arterctomy,abdominal aneurysm) , or major abdominal surgery .

Exclusion Criteria:

1. Hypersensitivity or knownallergy to amide local anesthetics
2. Pre-existing neurological deficit/peripheral neuropathy and Coagulation disorders.
3. Local infection at the site of block and at the planned cannulation site.
4. peripheral occlusive vascular disease, surgery for vascular injury or thromboembolic phenomena, cervical rib, and conditions associated with obstruction to arterial or venous flow.
5. Emergency operations and occlusion of the ipsilateral ulnar artery
6. patients on vasopressors and radial artery cannula removal before 24 hours postoperative.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The time to successful radial arterial cannulation | It will be measured from the initial needle penetration through the skin to removal of the metal needle and continuation of a flash of arterial blood in seconds at base line (15 minutes )before surgery
  It is measured from the initial needle penetration through the skin to removal of the metal needle and continuation of a flash of arterial blood in seconds

SECONDARY OUTCOMES:
Incidence of post cannulation complication such as arterial spasm , ischemia ,thrombosis and hematoma formation in the first 24 hours postoperative | It will be measured in the first 24 hours postoperative
  arterial spasm , ischemia ,thrombosis and hematoma formation

CONTACTS AND LOCATIONS:
Overall Officials: Amr ahmed abdel kader, lecturer, Study Director — Anesthesia department , Cairo university
Locations (2):
- Egypt (2):
  - Kasr Al Ainy, Cairo
  - Kasr Alainy, Cairo University, Cairo